CLINICAL TRIAL: NCT03441178
Title: A Prospective, Multi-Center Evaluation of the ENSEAL X1 Large Jaw Tissue Sealer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG-17-001
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Colectomy; Gynecological; Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Colectomy/Gynecological/Thoracic (Experimental): Any colectomy/gynecological/thoracic procedure where ENSEAL X1 is used for transecting and sealing vessels according to instructions for use.
  Interventions: Device: ENSEAL X1

INTERVENTIONS:
Device: ENSEAL X1 — ENSEAL X1 is used for transecting and sealing vessels according to instructions for use.

SUMMARY:
This prospective, single-arm, multi-center, evaluation will collect clinical data in a post-market setting. The three types of procedures studied will be colectomy, gynecological, and thoracic. Investigators will perform each procedure using the device in compliance with their standard surgical approach and the ENSEAL X1 instructions for use.

DETAILED DESCRIPTION:
The primary objective of this study is to prospectively generate device specific clinical data related to hemostasis in a post-market setting using the ENSEAL X1 per its instructions for use. There will be no blinding or planned interim analysis in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Elective procedure (colectomy, gynecological, or thoracic) where at least one vessel is planned to be transected by the ENSEAL X1 device per its instructions for use;
2. Willingness to give consent and comply with all study-related evaluations and treatment schedule; and
3. At least 18 years of age.

Exclusion Criteria:

1. Physical or psychological condition which would impair study participation; or
2. Enrollment in a concurrent clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Robb, MD, Principal Investigator — Indiana University
Locations (6):
- Indiana University, Indianapolis, Indiana, United States
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Planned on 100 enrolled but 101 was enrolled due to timing and study closure.
Groups:
- Colectomy; Thoracic: Any thoracic procedure where ENSEAL X1 is used for transecting and sealing vessels according to instructions for use.
- Gynecological: Any gynecological procedure where ENSEAL X1 is used for transecting and sealing vessels according to instructions for use.
Period: Overall Study
Arm/Group | Colectomy | Gynecological | Thoracic
Started | 36 | 44 | 21
Completed | 36 | 43 | 20
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- ENSEAL X1 Large Jaw Tissue Sealer: Use of the ENSEAL X1 Large Jaw Tissue Sealer
Arm/Group | ENSEAL X1 Large Jaw Tissue Sealer
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 96
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Vessels Where Hemostasis (<= Grade 3) is Achieved Using ENSEAL X1
Description: * Grade 1: no bleeding at transection site;
  * Grade 2: minor bleeding at transection site, no intervention needed;
  * Grade 3: minor bleeding at transection site, mild intervention needed, use of monopolar device and/or touch-ups with ENSEAL X1;
  * Grade 4: significant bleeding (e.g., pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or ligation with additional hemostatic products (e.g., hemoclips, staples, sutures, fibrin sealants, other advanced energy products).
Time Frame: Intraoperative, after vessel has been transected
Measure: Number (95% Confidence Interval); unit: Percentage of Vessels
Units Other Than Participants: Vessels Transected
Groups:
- Total: Any colectomy, gynecological or thoracic procedure where ENSEAL X1 is used for transecting and sealing vessels according to instructions for use.
Arm/Group | Colectomy | Gynecological | Thoracic | Total
Number analyzed (Participants) | 36 | 44 | 21 | 101
Number analyzed (Vessels Transected) | 68 | 156 | 90 | 314
Percentage of Vessels | 100.0 [94.7 to 100.0] | 94.2 [89.3 to 97.3] | 96.7 [90.6 to 99.3] | 96.2 [93.4 to 98.0]

2. Secondary Outcome: Hemostasis Grading Assessment for Each Vessel Transection
Description: as for outcome 1
Time Frame: Intraoperative, after vessel has been transected
Measure: Count of Units; unit: Vessels Transected
Units Other Than Participants: Vessels Transected
Arm/Group | Colectomy | Gynecological | Thoracic | Total
Number analyzed (Participants) | 36 | 44 | 21 | 101
Number analyzed (Vessels Transected) | 68 | 156 | 90 | 314
Vessels Transected
  Grade 1 | 63 | 126 | 81 | 270
  Grade 2 | 4 | 14 | 3 | 21
  Grade 3 | 1 | 7 | 3 | 11
  Grade 4 | 0 | 9 | 3 | 12

3. Secondary Outcome: Number of Grade 3 Vessels Needing ENSEAL X1 Touch-up
Description: as for outcome 1
Time Frame: Intraoperative, after vessel has been transected
Measure: Number; unit: Vessels Transected
Units Other Than Participants: Grade 3 Vessels
Arm/Group | Colectomy | Gynecological | Thoracic | Total
Number analyzed (Participants) | 36 | 44 | 21 | 101
Number analyzed (Grade 3 Vessels) | 1 | 7 | 3 | 11
Vessels Transected | 0 | 7 | 1 | 8

4. Secondary Outcome: Number of Hemostasis Grade 4 Transections and Hemostatic Interventions Used
Description: as for outcome 1
Time Frame: Intraoperative, after vessel has been transected
Population: There were no Grade 4 vessels seen in the colectomy procedures.
Measure: Number; unit: Vessels Transected
Units Other Than Participants: Grade 4 Vessels
Arm/Group | Gynecological | Thoracic | Total
Number analyzed (Participants) | 44 | 21 | 101
Number analyzed (Grade 4 Vessels) | 9 | 3 | 12
Vessels Transected
  Left uterine artery and vein (suture) | 2 | 0 | 2
  Left uterine artery (suture) | 2 | 0 | 2
  Right uterine artery (suture) | 4 | 0 | 4
  Right ovarian artery (suture) | 1 | 0 | 1
  Short gastric (suture -1; hemoclip -1) | 0 | 2 | 2
  Gastroepiploic (suture) | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: 4 Weeks Post Procedure
Arm/Group | ENSEAL X1 Large Jaw Tissue Sealer
All-Cause Mortality (participants affected / at risk) | 1/101
Serious Adverse Events (participants affected / at risk) | 12/101
Other Adverse Events (participants affected / at risk) | 43/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENSEAL X1 Large Jaw Tissue Sealer (N=101)
Ileus paralytic (Gastrointestinal disorders) | 1
Empyema (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 3
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENSEAL X1 Large Jaw Tissue Sealer (N=101)
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Pain (General disorders) | 11
Pyrexia (General disorders) | 3
Procedural pain (Injury, poisoning and procedural complications) | 16
Procedural vomiting (Injury, poisoning and procedural complications) | 4
Anastomotic leak (Injury, poisoning and procedural complications) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03441178/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03441178/SAP_001.pdf